CLINICAL TRIAL: NCT02256696
Title: A Phase 2 Randomized, Open-Label Trial of PA-824-Containing Regimens Versus Standard Treatment for Drug-Sensitive Sputum Smear-Positive Pulmonary Tuberculosis
Brief Title: Assessing PA-824 for Tuberculosis (the APT Trial)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: University of Cape Town (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00093014; #FD-R-004794-01 (Other: Office of Orphan Products Development (OOPD))
Record Dates: First submitted 2014-09-25; First posted 2014-10-06 (Estimated); Results first posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-05

CONDITIONS: Pulmonary Tuberculosis
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — pretomanid; Rifampin; Rifabutin; Pyrazinamide; Ethambutol; Isoniazid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): PA-824 200 mg once daily (QD),Rifampin 600 mg once daily, Isoniazid 5 mg/kg once daily, Pyrazinamide 25 mg/kg once daily x 8 weeks, then PA-824 200 mg once daily, Rifampin 600 mg once daily, Isoniazid 5 mg/kg once daily x 4 weeks
  Interventions: Drug: PA-824; Drug: Rifampin; Drug: Pyrazinamide; Drug: Isoniazid
- Arm 2 (Experimental): PA-824 200 mg once daily,Rifabutin 300 mg once daily , Isoniazid 5 mg/kg once daily, Pyrazinamide 25 mg/kg once daily x 8 weeks, then PA-824 200 mg once daily, Rifabutin 300 mg once daily, Isoniazid 5 mg/kg once daily x 4 weeks
  Interventions: Drug: PA-824; Drug: Rifabutin; Drug: Pyrazinamide; Drug: Isoniazid
- Arm 3 (Active Comparator): Rifampin 600 mg once daily, Ethambutol 15mg/kg once daily, Isoniazid 5 mg/kg once daily, Pyrazinamide 25 mg/kg once daily x 8 weeks, then Rifampin 600 mg once daily, Isoniazid 5 mg/kg once daily x 4 weeks
  Interventions: Drug: Rifampin; Drug: Pyrazinamide; Drug: Ethambutol; Drug: Isoniazid

INTERVENTIONS:
Drug: PA-824 — 200 mg QD
  Other Names: Pretomanid
  Arms: Arm 1; Arm 2
Drug: Rifampin — 600 mg QD
  Arms: Arm 1; Arm 3
Drug: Rifabutin — 300 mg QD
  Arms: Arm 2
Drug: Pyrazinamide — 25mg/kg QD
Drug: Ethambutol — 15mg/kg QD
  Arms: Arm 3
Drug: Isoniazid — 300 mg QD

SUMMARY:
Assess the mycobactericidal activity of PA-824 (given at 200 mg daily) when added to first-line tuberculosis (TB) treatment (isoniazid, pyrazinamide, and a rifamycin antibiotic) over 12 weeks of treatment. Funding Source - FDA Office of Orphan Products Development (OOPD)

DETAILED DESCRIPTION:
Phase IIB, 12-week, open-label, single-site, randomized clinical trial with three treatment groups. Patients with drug-sensitive TB will all receive once daily isoniazid and pyrazinamide for 8 weeks followed by 4 weeks of daily isoniazid. In addition, Arm 1 participants will receive PA-824 200 mg daily and rifampin 600 mg daily for 12 weeks. Arm 2 participants will receive PA-824 200 mg daily and rifabutin 300 mg daily for 12 weeks. Arm 3 participants (control group) will receive rifampin for 12 weeks and ethambutol for 8 weeks. Patients will be screened within 1 week of TB diagnosis, will receive 12 weeks of study treatment and will return for follow-up visits at 4, 12, and 36 weeks after study treatment completion. All patients will be referred to the local TB treatment program after completion of study treatment to finish their 24-week TB treatment course.

ELIGIBILITY:
Inclusion Criteria:

1. Suspected pulmonary tuberculosis with acid-fast bacilli in a stained smear of expectorated sputum or Gene Xpert positive sputum sample. Patients having extra-pulmonary manifestations of tuberculosis, in addition to smear-positive pulmonary disease, are eligible for enrollment.
2. Age > 18 years
3. . Weight ≥ 40 kg and ≤ 80 kg
4. Karnofsky score of at least 60 (requires occasional assistance but is able to care for most of his/her needs)
5. . Signed informed consent
6. . HIV negative, or positive with CD4 ≥350 cells/cu mm and not currently taking or planning to take combination antiretroviral therapy for HIV during the study.
7. Ability to adhere with study follow-up

8 Agrees to adhere to contraceptive requirements

-

Exclusion Criteria:

1. Pregnant or breast-feeding
2. Known intolerance or allergy to any of the study drugs
3. Concomitant disorders or conditions for which isoniazid, rifampin, rifabutin, pyrazinamide, or ethambutol is contraindicated. These include severe hepatic damage, acute liver disease of any cause, allergy to the drug, and acute uncontrolled gouty arthritis.
4. Current or planned therapy, during the intensive phase of TB therapy with cyclosporine or tacrolimus, which have unacceptable interactions with rifamycins.
5. Any medical or psychosocial condition, which, in the view of the study investigator, makes study participation inadvisable.
6. Pulmonary silicosis
7. Central nervous system TB
8. ECG at screening with corrected QT interval (QTc) (Fridericia correction) interval >450 ms or any clinically-significant, in the opinion of the investigator, ECG abnormality
9. History and/or presence (or evidence) of neuropathy or epilepsy.
10. History of lens opacity or evidence of lens opacity on slit lamp ophthalmologic examination with a value of 1.0 or higher on age-related eye disease scale 2 (AREDS2) Clinical Lens Opacity Classification and Grading System scale.
11. Infection with an isolate known to be resistant to a first-line TB drug (for example, patients with Gene Xpert screening through the local TB program with results suggesting resistance to rifampin)
12. Laboratory parameters done at, or 14 days prior to, screening (with results available for review by study personnel) demonstrating any of the following:

    * Serum alanine aminotransferase (ALT) activity > 3 times the upper limit of normal
    * Serum total bilirubin level > 2 times the upper limit of normal
    * Serum creatinine greater than the upper limit of normal
    * Hemoglobin level less than 7.0 g/dL
    * Platelet count less than 100,000/mm3
    * Positive pregnancy test (women of childbearing potential)
13. More than five days of treatment directed against active tuberculosis in the past 6 months -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2015-04-29 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly E Dooley, MD PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- University of Cape Town Lung Institute, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: Yes
This plan is in process, to be finalized prior to the end of recruitment.
Time Frame: Within one year of reaching recruitment goals.
Access Criteria: This plan is in process, to be finalized prior to the end of recruitment.

REFERENCES:
- [Derived] Dooley KE, Hendricks B, Gupte N, Barnes G, Narunsky K, Whitelaw C, Smit T, Ignatius EH, Friedman A, Dorman SE, Dawson R; Assessing Pretomanid for Tuberculosis (APT) Study Team. Assessing Pretomanid for Tuberculosis (APT), a Randomized Phase 2 Trial of Pretomanid-Containing Regimens for Drug-Sensitive Tuberculosis: 12-Week Results. Am J Respir Crit Care Med. 2023 Apr 1;207(7):929-935. doi: 10.1164/rccm.202208-1475OC. PMID 36455068
- [Derived] Ignatius EH, Abdelwahab MT, Hendricks B, Gupte N, Narunsky K, Wiesner L, Barnes G, Dawson R, Dooley KE, Denti P. Pretomanid Pharmacokinetics in the Presence of Rifamycins: Interim Results from a Randomized Trial among Patients with Tuberculosis. Antimicrob Agents Chemother. 2021 Jan 20;65(2):e01196-20. doi: 10.1128/AAC.01196-20. Print 2021 Jan 20. PMID 33229425

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1 | Arm 2 | Arm 3
Started | 56 | 53 | 48
Completed | 53 | 50 | 47
Not Completed | 3 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Total
Number analyzed (Participants) | 56 | 53 | 48 | 157
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 32 [25 to 39] | 30 [23 to 35] | 31 [23 to 40] | 31 [23 to 39]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 17 | 9 | 39
  Male | 43 | 36 | 39 | 118
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 38 | 35 | 29 | 102
  Colored | 18 | 18 | 18 | 54
  Other | 0 | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 56 | 53 | 48 | 157
  >=65 years | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to Sputum Culture Conversion on Liquid Medium
Description: The time (days) it takes for the sputum to convert from positive to negative.
Time Frame: 12 weeks
Population: Adult (> 18 years) drug sensitive pulmonary TB patients with weight 40 - 80 kg, HIV Negative or Positive with CD4 > 350, not on antiretroviral therapy (ART)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 53 | 50 | 47
days
  Time to culture conversion (mITT) | 42 [21 to 56] | 28 [21 to 42] | 56 [42 to 70]
  Time to culture conversion (per protocol): number analyzed (Participants) | 51 | 43 | 47
  Time to culture conversion (per protocol) | 42 [21 to 56] | 28 [21 to 42] | 56 [42 to 70]
Statistical Analysis 1: Comparison: Arm 1 vs Arm 3; modified intention to treat (mITT) analysis; Test type: Superiority; p = 0.10, Regression, Cox; adjusted for age and sex at birth; Hazard Ratio (HR) = 1.41, 95% CI 2-sided [0.93 to 2.12]
Statistical Analysis 2: Comparison: Arm 2 vs Arm 3; mITT analysis; Test type: Superiority; p = 0.003, Regression, Cox; adjusted for age and sex at birth; Hazard Ratio (HR) = 1.89, 95% CI 2-sided [1.24 to 2.87]
Statistical Analysis 3: Comparison: Arm 1 vs Arm 3; per protocol; Test type: Superiority; p = 0.09, Regression, Cox; adjusted for age and sex at birth; Hazard Ratio (HR) = 1.43, 95% CI 2-sided [0.95 to 2.15]
Statistical Analysis 4: Comparison: Arm 2 vs Arm 3; per protocol; Test type: Superiority; p = 0.005, Regression, Cox; adjusted for age and sex at birth; Hazard Ratio (HR) = 1.87, 95% CI 2-sided [1.21 to 2.89]

2. Primary Outcome: Number of Participants With Grade 3 or Higher Adverse Events
Description: Any Grade 3 event according to the Division of AIDS (DAIDS) toxicity table
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 56 | 53 | 48
Participants | 3 | 6 | 2

3. Secondary Outcome: Number of Participants With Permanent Discontinuation of Assigned Study Regimen
Description: If it is in the best interest of a participant to stop the study regimen for any reason
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 56 | 53 | 48
Participants | 2 | 7 | 0

4. Secondary Outcome: Time to Culture Conversion on Solid Medium
Description: The time (days) it takes for the sputum to convert form positive to negative on solid medium
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 56 | 53 | 48
days
  Time to conversion on solid culture (mITT) | 28 [14 to 42] | 21 [14 to 28] | 42 [21 to 56]
  Time to conversion on solid culture (per protocol) | 28 [14 to 42] | 21 [14 to 28] | 42 [21 to 56]
Statistical Analysis 1: Comparison: Arm 1 vs Arm 3; mITT analysis; Test type: Superiority; p = 0.02, Regression, Cox; adjusted for age and sex at birth; Hazard Ratio (HR) = 1.61, 95% CI 2-sided [1.07 to 2.44]
Statistical Analysis 2: Comparison: Arm 2 vs Arm 3; mITT analysis; Test type: Superiority; p = 0.006, Regression, Cox; adjusted for age and sex at birth; Hazard Ratio (HR) = 1.80, 95% CI 2-sided [1.18 to 2.75]
Statistical Analysis 3: Comparison: Arm 1 vs Arm 3; per protocol analysis; Test type: Superiority; p = 0.03, Regression, Cox; adjusted for age and sex at birth; Hazard Ratio (HR) = 1.60, 95% CI 2-sided [1.05 to 2.42]
Statistical Analysis 4: Comparison: Arm 2 vs Arm 3; per protocol analysis; Test type: Superiority; p = 0.007, Regression, Cox; adjusted for age and sex at birth; Hazard Ratio (HR) = 1.84, 95% CI 2-sided [1.18 to 2.85]

5. Secondary Outcome: Percentage of Participants With Sputum Culture Conversion by 8 Weeks of Treatment
Description: Percentage of participants whose sputum converts from positive to negative at Week 8 time point, on solid and liquid media.
Time Frame: 8 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 56 | 53 | 48
percentage of participants
  Liquid media | 79 | 89 | 69
  Solid media | 98 | 100 | 96

6. Secondary Outcome: Steady State Pharmacokinetics (PK) (AUC) of PA-824 When Given With Rifampin or Rifabutin
Description: AUC of PA-824 when given with either rifampicin or rifabutin to determine steady state Pharmacokinetics (PK) of PA-824.
Time Frame: pre-dose and 1, 2, 5, 8, and 24 hours post-dose on Day 14
Population: This outcome was not assessed in Arm 3, because no participants received PA-824 in Arm 3.
Measure: Mean (Standard Deviation); unit: mg*h/L
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 56 | 53
mg*h/L | 31.91 (9.87) | 59.05 (13.30)

7. Secondary Outcome: PK (Cmax) of PA-824 at 200 mg Once Daily With Rifampin or Rifabutin-containing Treatment
Description: The Pharmacokinetic results (Cmax) of the study drug when given with a rifampin or a rifabutin.
Time Frame: pre-dose and 1, 2, 5, 8, and 24 hours post-dose on Day 14
Population: This outcome was not assessed in Arm 3, because no participants received PA-824 in Arm 3.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 56 | 53
mg/L | 2.03 (0.51) | 2.69 (0.82)

8. Secondary Outcome: Relationship Between PA-824 Exposure (AUC) and Rate of Change in Time to Positivity (TTP) Over 12 Weeks
Description: Relationship between PA-824 exposure (AUC) and rate of change in TTP over 12 weeks, using non-linear mixed effects modeling. The data is reported as percentage increase in TTP per 10 unit increase in PA-824 AUC (% increase/10 unit increase PA-824 AUC).
Time Frame: 12 weeks
Population: This outcome was measured among all participants receiving study drug (PA-824), as one group.
Measure: Number (95% Confidence Interval); unit: % increase/10 unit increase PA-824 AUC
Groups:
- Arms 1 and 2 (Pretomanid-containing Arms): This is a combined measure drawn from both arms 1 and 2, in which participants received PA-824 (pretomanid)
Arm/Group | Arms 1 and 2 (Pretomanid-containing Arms)
Number analyzed (Participants) | 109
% increase/10 unit increase PA-824 AUC | 9.4 [4.4 to 15.5]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Arm 1 | Arm 2 | Arm 3
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/53 | 0/48
Serious Adverse Events (participants affected / at risk) | 3/56 | 4/53 | 0/48
Other Adverse Events (participants affected / at risk) | 3/56 | 3/53 | 2/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (N=56) | Arm 2 (N=53) | Arm 3 (N=48)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleuritic chest pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Increased liver enzymes (Hepatobiliary disorders) | 0 | 3 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (N=56) | Arm 2 (N=53) | Arm 3 (N=48)
Low hemoglobin (Blood and lymphatic system disorders) | 1 | 2 | 1
Drug induced liver injury (Hepatobiliary disorders) | 1 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Increased blood pressure (Cardiac disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-02-07): https://cdn.clinicaltrials.gov/large-docs/96/NCT02256696/Prot_SAP_000.pdf
  • Informed Consent Form (2020-05-28): https://cdn.clinicaltrials.gov/large-docs/96/NCT02256696/ICF_001.pdf